CLINICAL TRIAL: NCT01288586
Title: Post-Approval Study to Investigate the Long Term (8 Year) Survivorship of Scandinavian Total Ankle Replacement (STAR) Ankle Among Continued Access Study Patients
Brief Title: Post-Approval Study to Investigate the Long Term (8 Year) Survivorship of STAR Ankle Among Continued Access Study Patients
Acronym: STAR 8
Status: Completed | Type: Observational
Sponsor: Stryker Trauma and Extremities (Industry)
Responsible Party: Sponsor
Other Study IDs: STAR 8 Year; NCT00586144 (obsolete NCT alias); NCT00586768 (obsolete NCT alias)
Record Dates: First submitted 2010-11-04; First posted 2011-02-02 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Primary Arthrosis
Keywords: Post Traumatic Arthritis; Rheumatoid Arthritis; Osteoarthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Device: Scandinavian Total Ankle Replacement System (STAR Ankle)
  Interventions: Device: Scandinavian Total Ankle Replacement System (STAR Ankle)

INTERVENTIONS:
Device: Scandinavian Total Ankle Replacement System (STAR Ankle) — Total Ankle Replacement
  Other Names: STAR

SUMMARY:
The purpose of this study is to examine the long term survivorship of the Scandinavian Total Ankle Replacement (STAR). Specifically, this study focuses on the revision and/or removal rate of any component of the STAR ankle.

ELIGIBILITY:
The study population consists of all living subjects who participated in the continued access arm of the IDE clinical trial.

Inclusion Criteria:

* Only patients that participated in the continued access study make up the patient cohort for this long-term follow-up study.
* Willing and able to give informed consent.

Exclusion Criteria:

* Subjects who were withdrawn or withdrew consent to participate in the investigation
* Subjects who do not consent to participate in long-term or provide personal contact information to the sponsor(solely for the purposes of tracking subjects to help ensure follow-up compliance)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of all living subjects who participated in the continued access study.
Sampling Method: Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2009-10-05 (Actual); Primary Completion 2016-11-14 (Actual); Study Completion 2016-11-14 (Actual)

PRIMARY OUTCOMES:
The primary objective for this study is to examine the long-term survivorship of the STAR Ankle | 8 year
  Obtain information on the revision and removal rate for the STAR Ankle over time.

SECONDARY OUTCOMES:
American Orthopaedic Foot and Ankle Society questionnaire will be used to evaluate and monitor the progress of patients following foot and ankle surgery. | 8 year

CONTACTS AND LOCATIONS:
Overall Officials: Richard Jay, DPM, Study Director — Stryker Nordic
Locations (5):
- United States (5):
  - Oakland Bone & Joint Specialists, Oakland, California
  - Foundations of Orthopedic Research and Education, Temple Terrace, Florida
  - St. Alphonsus Medical Group, Coughlin Foot & Ankle Clinic, Boise, Idaho
  - Kansas University Medical Center, Kansas City, Kansas
  - Duke University, Durham, North Carolina